CLINICAL TRIAL: NCT07021352
Title: Effects of Auricular Acupuncture on Emotional Distress in Service Members and Veterans With Posttraumatic Stress Disorder
Brief Title: Auricular Acupuncture on Emotional Distress in Service Members and Veterans With PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jane J. Abanes, Assistant Professor, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSNRP N25D272IR
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: PTSD and Substance Use Disorder; Emotional Distress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear acupuncture plus mindfulness therapy (Experimental): Arm A (Ear Acupuncture plus Mindfulness): Participants will receive bilateral NADA ear acupuncture protocol treatment for a one-time insertion in addition to the weekly mindfulness therapy received by participants. The NADA consists of 5 ear acupuncture points inserted bilaterally: shen men, sympathetic, kidney, liver, and lung. Sterile, semi-permanent acupuncture needles (2mm) will be inserted into the participant's ear and left in place until they naturally fall out, typically within 3-7 days. This group will also receive mindfulness weekly for 30 minutes each session via the MS Teams platform.
  Interventions: Procedure: Ear acupuncture; Behavioral: Mindfulness therapy
- Mindfulness Therapy Only (Active Comparator): Arm B (Mindfulness only): The mindfulness-only group will receive mindfulness therapy weekly. Participants in arm B will receive virtual mindfulness weekly for 30 minutes each session via the MS Teams platform.
  Interventions: Behavioral: Mindfulness therapy

INTERVENTIONS:
Procedure: Ear acupuncture — Ear Acupuncture: Participants will receive bilateral NADA ear acupuncture protocol treatment for a one-time insertion in addition to the weekly mindfulness therapy received by participants. The NADA consists of 5 ear acupuncture points inserted bilaterally: shen men, sympathetic, kidney, liver, and lung. Sterile, semi-permanent acupuncture needles (2mm) will be inserted into the participant's ear and left in place until they naturally fall out, typically within 3-7 days.
  Arms: Ear acupuncture plus mindfulness therapy
Behavioral: Mindfulness therapy — Mindfulness: Participants will receive virtual mindfulness therapy weekly for 30 minutes each session via the MS Teams platform.

SUMMARY:
Emotional distress (ED) refers to a state of mental suffering that significantly impairs an individual's ability to cope, often leading to a decline in overall well-being. In military contexts, ED is a prevalent concern due to the unique and demanding challenges faced by military personnel both in combat zones and during peacetime. The primary objective of this study is to assess the efficacy of integrating ear acupuncture with mindfulness therapy in mitigating ED and alleviating post-traumatic stress disorder (PTSD) symptoms among military personnel. The study will examine the effects of auricular acupuncture (AA) and mindfulness therapy (MT) on ED in military personnel with PTSD. The NADA ear acupuncture protocol will be administered using acupuncture semi-permanent (ASP), sterile needles placed in the bilateral ears, which will remain in place until they naturally fall out. Mindfulness therapy will incorporate relaxation techniques, such as yoga and controlled breathing exercises, specifically designed to alleviate ED. A mixed-methods approach, integrating both quantitative and qualitative methods, will be employed concurrently to evaluate the interventions' effectiveness and to explore the participants' perceived benefits. Specific Aim 1: To evaluate the effectiveness and perceived benefits of the National Acupuncture Detoxification Association (NADA) ear acupuncture protocol as an adjunct therapy to brief mindfulness therapy for reducing emotional distress in service members and veterans with PTSD. Specific Aim 2: To examine the effectiveness of NADA as an adjunct therapy to brief mindfulness therapy in improving sleep disturbances, alcohol use, and pain in service members and veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service member and veterans
* A score of 14 or above on the abbreviated PCL 6-item
* A score of 24 or above on the EDS
* Agrees to participate in mindfulness therapy
* Able to provide informed consent

Exclusion Criteria:

- Has had mindfulness therapy received from a healthcare provider in the past month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Emotional Distress - Anger Short Form 8a | Baseline, post 2-week intervention, post 4-week intervention
  Minimum value= 5, Maximum value = 40; higher scores mean worse outcome

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for Diagnostic Statistical Manual-5 | Baseline, post 2-week intervention, post 4-week intervention
  Minimum value = 0, Maximum value = 80, higher scores mean worse outcome
Insomnia Severity Index | Baseline, post 2-week intervention, post 4-week intervention
  Minimum value= 0, Maximum value = 28; higher scores mean worse outcome
Alcohol Use Disorders Identification Test | Baseline, post 2-week intervention, post 4-week intervention
  Minimum value= 0, Maximum value = 40; higher scores mean worse outcome
Numeric Rating Scale | Baseline, post 2-week intervention, post 4-week intervention
  Minimum value= 0, Maximum value = 10; higher scores mean worse outcome

IPD SHARING:
Plan to Share IPD: Undecided